CLINICAL TRIAL: NCT00196222
Title: European Multicenter Study RF Versus Cryo in AVNRT: A Randomized Study Comparing Cryo-Energy vs. Radiofrequency-Energy Ablation Technique for AV Nodal Reentry Tachycardia (AVNRT)
Brief Title: European Multicenter Study Radiofrequency (RF) Versus Cryo in Atrioventricular Nodal Reentry Tachycardia (AVNRT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: CryoCath Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. C00403
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Atrioventricular Nodal Reentry Tachycardia
MeSH Terms: conditions — Tachycardia, Atrioventricular Nodal Reentry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): RF ablation/modulation of the slow pathway in AV nodal reentrant tachycardia
  Interventions: Procedure: RF-ablation
- 2 (Experimental): cryo energy ablation/modulation of the slow pathway in AV nodal reentrant tachycardia
  Interventions: Procedure: cryo ablation

INTERVENTIONS:
Procedure: RF-ablation — RF ablation/modulation of the slow pathway in AV nodal reentrant tachycardia
  Arms: 1
Procedure: cryo ablation — Cryo ablation/modulation of the slow pathway in AV nodal reentrant tachycardia
  Arms: 2

SUMMARY:
In this randomized study, two energy sources for the ablation of AV nodal reentry tachycardia are compared: The standard technique of radiofrequency energy delivery is compared with the new approach of cryo-energy application.

DETAILED DESCRIPTION:
The ablation of AV nodal reentry tachycardia with radiofrequency (RF) energy delivering catheters is a standard procedure and in experienced EP laboratories, the safety and efficacy of this approach is very high.

However, the potential complication of higher degree AV conduction block, requiring in some instances implantation of a pacemaker, is a major drawback of this approach.

We want to compare in this randomized study the safety and efficacy of standard RF ablation with the cryo-ablation technique. This relatively new technique is thought to offer more safety concerning higher degree AV conduction block.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years old
* Clinical diagnosis of AVNRT (ECG/patients history)
* Electrophysiologically confirmed (invasively assessed) diagnosis of AVNRT
* Written informed consent

Exclusion Criteria:

* Prior ablation for AVNRT
* Congenital heart disease interfering with the ablation method
* Prior cardiac surgery
* Medical or psychiatric disorder interfering with study protocol or data acquisition
* Exclusion of the patient by the study investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2003-03; Primary Completion 2008-11 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Combined endpoint of safety and efficacy of cryo ablation compared with RF ablation for procedure and 6 months follow-up data. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Claus Schmitt, MD, Study Chair — Deutsches Herzzentrum Muenchen; Bernhard Zrenner, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (10):
- Germany (10):
  - Kerckhoffklinik GmbH EPU, Bad Nauheim
  - Charite Berlin Virchow - Klinikum Med. Klinik, Berlin
  - Universitaetsklinikum Bonn Med. Klinik II, Bonn
  - Evangelisches Krankenhaus Duesseldorf Kardiologie, Düsseldorf
  - Universitaetsklinikum Giessen EPU, Giessen
  - Klinikum Luedenscheid Kardiologie, Lüdenscheid
  - Klinikum der Stadt Mannheim Med. Klinik I, Mannheim
  - Deutsches Herzzentrum Muenchen, Munich
  - Universitaetsklinikum Tuebingen Med. Klinik/Abt.III, Tübingen
  - Universitaetsklinikum Ulm Innere Med. II, Ulm

REFERENCES:
- [Result] Deisenhofer I, Zrenner B, Yin YH, Pitschner HF, Kuniss M, Grossmann G, Stiller S, Luik A, Veltmann C, Frank J, Linner J, Estner HL, Pflaumer A, Wu J, von Bary C, Ucer E, Reents T, Tzeis S, Fichtner S, Kathan S, Karch MR, Jilek C, Ammar S, Kolb C, Liu ZC, Haller B, Schmitt C, Hessling G. Cryoablation versus radiofrequency energy for the ablation of atrioventricular nodal reentrant tachycardia (the CYRANO Study): results from a large multicenter prospective randomized trial. Circulation. 2010 Nov 30;122(22):2239-45. doi: 10.1161/CIRCULATIONAHA.110.970350. Epub 2010 Nov 15. PMID 21098435